CLINICAL TRIAL: NCT04993274
Title: Sensitivity of Quantitative Motor Performance Measures in Multiple Sclerosis - a Prospective Cohort Study Over Two Years Using Microsoft Kinect
Brief Title: Sensitivity of Motor Assessment in MS - a Prospective Cohort Study
Acronym: MOTOSENS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Friedemann Paul (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Friedemann Paul, Direktor ECRC, Leiter AG Klinische Neuroimmunologie, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: EA1/240/18
Record Dates: First submitted 2021-03-09; First posted 2021-08-06 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Secondary Progressive; Multiple Sclerosis, Chronic Progressive
Keywords: multiple sclerosis; gait; balance; postural control; progression; observational; assessment; motion capture
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PASS-MS — protocol using short motor tasks performed by the subject and recorded by a depth camera, motion analysis by visuo-perceptive computing

SUMMARY:
The study explores the application of marker-less motion analysis (visual-perceptive computing, VPC) using a consumer grade infrared and video camera (Microsoft Kinect) for clinical assessment in MS. It includes as the primary outcomes a short assessment battery of simple motor tasks (PASS-MS) that can be performed in front of the sensor after standard oral instructions given by the operator. For each task, the sensor data are transformed into a set of kinematic parameters that may be used as motor outcome reflecting specific neurological dysfunction. For validation against both clinical and patient-reported outcomes as well as MRI findings, we here prospectively investigate a large cohort of patients with multiple sclerosis. This will allow to determine the usefulness of the various kinematic parameters generated and to define a reduced set of the most meaningful parameters for potential use in future MS trials. Data on repeatability and benchmarks for clinically relevant change are essential to interpret test results and, more importantly, changes thereof. Further, this prospective study will yield estimates of progression rates that are required for planning future studies using this motion analysis tool and assessment battery as an outcome. The study is designed to obtain benchmarks for sensitivity and clinical responsiveness. Primary analysis aims to answer the question: Does the SMSW - Maximum Speed worsen with disease progression established as confirmed disability progression based on EDSS after 24 months (defined as 1 step increase in EDSS ≤ 5.5 and 0.5 step in EDSS > 5.5)?

DETAILED DESCRIPTION:
The study is designed as a prospective observational (non-interventional) single-center study performed at one center, Charité - Universitätsmedizin Berlin.

This study converges with prospective observational studies performed at our center. These studies started in 2011 with the objective to define determinants of progression in neuroimmunological disorders (CIS, MS, NMO).

The variables collected for this study were defined according to the study objective and comprise different markers of motor/mobility function, cognitive and affective function, fatigue and health-related quality of life. The primary outcome is a VPC-based assessment of locomotor function (PASS-MS SMSW-MaxS) as the diagnostic test under study. Secondary outcomes serve to cross-validate progression rates or as benchmarks of clinical progression to determine clinical relevance of change. Further, possible effects of cognitive and affective function on the primary outcome can be explored which is of high relevance for the interpretation of changes in the population of MS.

All assessments are performed at inclusion and after 12and 24 months.

Primary outcome:

PASS-MS kinematic parameters with Short Maximum Speed Walk - Speed (SMSW-MaxS) as primary outcome

Secondary outcomes:

* Clinical Examination
* Other kinematic parameters derived from PASS-MS
* Clinical Rating with EDSS and Multiple Sclerosis Functional Composite (MSFC) consisting of tests of walking capacity (T25FW), hand dexterity (9HPT), cognitive processing speed (SDMT) and visual acuity (Sloan charts)
* Cognitive testing (BRB-N)
* Patient-reported outcomes on global impression of change, MS-related impairment in walking (MSWS-12), hand function, occurrence of fatigue (FSMC), depressive symptoms (BDI-II) and health-related quality of life by MS-specific questionnaire (HAQUAMS)

A change in T25FW speed of at least 20% was found to be clinically meaningful for MS patients (Hobart 2013). In a previous study the investigators found SMSW average walking speed was slower in MS patients (1.6 ± 0.3 m/sec) than in HC (1.8 ± 0.4 m/sec) (Behrens 2014). Therefore, a similar average walking speed was assumed for the population under study at baseline (1.6 m/sec) and a decrease of 0.3 m/sec (corresponding to approximately 20%) as clinically meaningful. Moreover, based on previous reports, investigators assume a standard deviation in the changes of SMSW-MaxS of 0.4 m/sec (Behrens 2014). This results in an expected effect size of 0.75 for the change in SMSW-MaxS between baseline and 24 months follow-up in those with clinically confirmed disability progression. A sample size of N=16 patients will have a power of 80% to detect an effect size of 0.75 with a two-sided significance level of 0.05 and a t-test for dependent samples (nQuery Advisor 7.0).

Sample size estimation considered previous evidence on the proportion of patients who will show clinically confirmed disability progression throughout the observation period based on an EDSS change defined as 1 step increase in EDSS ≤ 5.5 and 0.5 step in EDSS > 5.5 within 24 months. Cutter et al. (1999) reported that 10% of their patients showed EDSS confirmed sustained change within 3 months and 40% showed a change to baseline in 1 year reported in MSFC, which also incorporates the T25FW. The investigators assume that at least 20 % of patients showing a confirmed sustained change in EDSS according to above definition within 24months to be a realistic scenario.

When considering an overall dropout rate of 10-20% (lost to follow-up), this would result in N=16 complete datasets when overall N=100 patients are included.

Patients should not have had an acute relapse up to 3 months before follow-up visit (12 and 24 months). To avoid dropout due to acute relapse the follow-up visit is extended to up to 3 months in case of acute relapse.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of multiple sclerosis (relapsing-remitting, secondary or primary chronic progressive)
* ability to perform PASS-MS short walking test (max. of 5 m distance) with no or only unilateral assistance (EDSS <6.5)
* written consent

Exclusion Criteria:

* Inability to understand/ follow test instructions for any reason
* Other cause of locomotor or balance dysfunction than MS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to include and follow-up 100 patients with a diagnosis of MS according to revised McDonald criteria including relapsing-remitting and progressive disease courses. The design as a single-center study implied that broad inclusion criteria (RRMS, SPMS, PPMS) should be used in order to obtain robust results. We therefore chose not to limit recruitment to progressive MS, which would have required a multi-center study. Still, we conceive the main results of our study - sensitivity and responsiveness - to be conferrable to progressive MS (yet not the progression rates).
  We restrict inclusion to those able to walk at least short distance with unilateral assistance according to the testing requirements of the primary outcome. We further include patients with any intervention for MS or other morbidity as long as this is not considered to affect balance or locomotor function. Type of MS treatment and comorbidities are documented at baseline and follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
change in PASS-MS kinematic parameter Short Maximum Speed Walk - Speed (SMSW-MaxS) | change from baseline value at 2 years
  walking speed calculated from short distance walking in the SMSW task

CONTACTS AND LOCATIONS:
Overall Officials: Friedemann Paul, Principal Investigator — Experimental and Clinical Research Center, Charité - Universitätsmedizin Berlin, Germany
Locations (1):
- Experimental and Clinical Research Center, Studienambulanz Neuroimmunologie am Standort NCRC, Campus Mitte,Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ellinghaus CA, Rohling HM, Dorsch EM, Sperber PS, Arsenova R, Buenrostro GS, Rekers S, Usnich T, Schindler P, Kroneberg D, Bellmann-Strobl J, Oertel FC, Brandt AU, Weygandt M, Paul F, Piper SK, Schmitz-Hubsch T. Anchor-based evaluation of digital motor biomarkers from a 2-year observation in 100 patients with multiple sclerosis. J Neurol. 2025 Dec 4;273(1):4. doi: 10.1007/s00415-025-13541-y. PMID 41342942